CLINICAL TRIAL: NCT06052449
Title: Assessing Social Determinants of Health to Increase Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro2023-0374
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: screening; social determinants of health; lung cancer screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social determinants of health screening (Experimental): Participants will receive a social determinants of health screening assessment and referral process in addition to the community-based lung cancer screening educational tool.
  Interventions: Behavioral: Social determinants of health screening assessment and referral process; Behavioral: Current practice - Community-based lunch cancer screening (LungTalk)
- Community-based lung cancer screening (Active Comparator): Participants will receive a community-based lung cancer screening educational tool.
  Interventions: Behavioral: Current practice - Community-based lunch cancer screening (LungTalk)

INTERVENTIONS:
Behavioral: Social determinants of health screening assessment and referral process — Unite Us is an electronic SDoH screening and referral tool assessing: (1) financial resource strain; (2) housing stability; (3) transportation needs; and (4) food insecurity. Upon completion, the Unite Us platform identifies a list of geographically-tailored resources to connect the individual in need. A staff member will administer the SDoH screening and referral tool, review the results with the participant, and use the geographically-tailored resources to make SDoH-related referrals.
  Arms: Social determinants of health screening
Behavioral: Current practice - Community-based lunch cancer screening (LungTalk) — The current practice during community events is to offer LungTalk. LungTalk is a novel theoretically grounded health educational tool that will be delivered via iPad and is an interactive computer-based program that includes audio, video and animation segments with scripts presented from a master content library in consideration of different ways people like to learn. Informed by our prior research, LungTalk tailors its content based on smoking status and perceived barriers. In prior work, LungTalk more than doubled LCS knowledge and health beliefs (p < 0.01), and was associated with a significant increase in deciding to screen for lung cancer compared to control group; OR 1.99; 95% Confidence Interval (CI), 1.03, 3.85, p = 0.03.

SUMMARY:
A multilevel lung screening intervention that pairs Social Determinants of Health (SDoH) screening and referral with a tailored health communication and decision support tool for lung screening has the potential to significantly impact lung screening uptake among at-risk individuals in the community, particularly among those who face barriers related to SDoH. In addition, findings will advance the understanding of effective strategies for improving lung screening and prevention efforts in non-traditional settings, with the ultimate goal of reducing the burden of lung cancer. As ways to support the realization of the public health benefit of lung cancer screening are considered, multiple strategies and venues to reach, and intervene, with screening-eligible is key.

The goal of this study is to compare the effectiveness of a community-based lung screening educational tool paired with a social determinants of health (SDoH) screening assessment and referral process compared to a community-based lung cancer screening (LCS) educational tool alone as part of community outreach activities to improve (a) LCS rates (primary outcome); (b) intention to screen; and (c) individual-level potential drivers of LCS (health literacy, mistrust, stigma, fatalism, knowledge, health beliefs). It is hypothesized that providing SDoH screening and referral will result in higher levels of LCS, forward movement of intention to screen, and improved individual-level drivers of LCS.

DETAILED DESCRIPTION:
The study will be a pilot randomized controlled trial (RCT) to compare primary (LCS uptake) and secondary outcomes (intent to screen, literacy, mistrust, stigma, fatalism, health beliefs) among LCS-eligible men and women in New Jersey community-based settings who receive a community-based LCS educational tool paired with a social determinants of health (SDoH) screening assessment and referral process (n=50) compared to a community-based LCS educational tool alone (n=50) as part of community outreach activities. All individuals who attend a community event are normally assessed for cancer risks and appropriate cancer screening education is provided. For those who are eligible for LCS, they will also be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years to 80 years
* Currently smoke or quit smoking within the past 15 years
* 20 pack-year smoking history
* Has never had lung cancer screening
* Able to provide informed consent
* Able to speak and understand English

Exclusion Criteria:

* Diagnosed with lung cancer
* Has a history of having a lung cancer screening scan
* Unable to speak and understand English

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Lung cancer screening uptake | 1 months post intervention
  Number of participants in the two groups that get screened (have a computed tomography (CT or CAT) scan)

SECONDARY OUTCOMES:
Health Literacy | Baseline
  Health Literacy will be measured using the 3-item health literacy scale ranging from 0 (low health literacy level) to 12 (high health literacy level)
Health Literacy | 1 months post intervention
  Health Literacy will be measured using the 3-item health literacy scale ranging from 0 (low health literacy level) to 12 (high health literacy level)
Medical Mistrust | Baseline
  Medical Mistrust will be measured with 5 items ranging from 5 (low mistrust) to 25 (high mistrust)
Medical Mistrust | 1 months post intervention
  Medical Mistrust will be measured with 5 items ranging from 5 (low mistrust) to 25 (high mistrust)
Perceived Smoking-Related Stigma | Baseline
  Perceived Smoking-Related Stigma will be measured using the 5-item smoking-related stigma subscale of the Cataldo Lung Cancer Stigma Scale ranging from 5 (low perceived stigma) to 25 (high perceived stigma)
Perceived Smoking-Related Stigma | 1 months post intervention
  Perceived Smoking-Related Stigma will be measured using the 5-item smoking-related stigma subscale of the Cataldo Lung Cancer Stigma Scale ranging from 5 (low perceived stigma) to 25 (high perceived stigma)
Lung Cancer Fatalism | Baseline
  Lung Cancer Fatalism will be measured with 11 items ranging from 0 (no fatalism) to 11 (high fatalism)
Lung Cancer Fatalism | 1 months post intervention
  Lung Cancer Fatalism will be measured with 11 items ranging from 0 (no fatalism) to 11 (high fatalism)
Knowledge of Lung Cancer and Lung Screening | Baseline
  Knowledge of Lung Cancer and Lung Screening will be assessed with a 7-item multidimensional scale used in our preliminary studies adapted from literature specific to lung cancer. Several aspects will be assessed, including knowledge of lung cancer, risk, and screening. Range of scores is 0 (no knowledge) to 7 (high level of knowledge).
Knowledge of Lung Cancer and Lung Screening | 1 months post intervention
  Knowledge of Lung Cancer and Lung Screening will be assessed with a 7-item multidimensional scale used in our preliminary studies adapted from literature specific to lung cancer. Several aspects will be assessed, including knowledge of lung cancer, risk, and screening. Range of scores is 0 (no knowledge) to 7 (high level of knowledge).
Perceived Barriers to Lung Cancer Screening Scale | Baseline
  Perceived Barriers to Lung Cancer Screening Scale will be used ranging from 17 (low perceived barriers to lung screening) to 68 (high perceived barriers to lung screening).
Perceived Barriers to Lung Cancer Screening Scale | 1 months post intervention
  Perceived Barriers to Lung Cancer Screening Scale will be used ranging from 17 (low perceived barriers to lung screening) to 68 (high perceived barriers to lung screening).
Stage of Adoption for Decision-Making About Lung Screening | Baseline
  Stage of Adoption for Decision-Making About Lung Screening will be assessed with an algorithm of questions used in our prior studies assessing the 7 stages (unaware, aware but unengaged, undecided, decided not to act, decided to act, action, and maintenance). This will allow us to assess intent if someone has "decided to act".
Stage of Adoption for Decision-Making About Lung Screening | 1 months post intervention
  Stage of Adoption for Decision-Making About Lung Screening will be assessed with an algorithm of questions used in our prior studies assessing the 7 stages (unaware, aware but unengaged, undecided, decided not to act, decided to act, action, and maintenance). This will allow us to assess intent if someone has "decided to act".

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carter-Bawa, PhD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Meridian Health - Center for Discovery and Innovation, Nutley, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cancer Facts & Figures 2023. American Cancer Society, Inc.; 2022. https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/2023-cancer-facts-figures.html
- [Background] Pettit N, Ceppa D, Monahan P. Low Rates of Lung and Colorectal Cancer Screening Uptake Among a Safety-net Emergency Department Population. West J Emerg Med. 2022 Aug 11;23(5):739-745. doi: 10.5811/westjem.2022.5.55351. PMID 36205665
- [Background] Carter-Harris L, Ceppa DP, Hanna N, Rawl SM. Lung cancer screening: what do long-term smokers know and believe? Health Expect. 2017 Feb;20(1):59-68. doi: 10.1111/hex.12433. Epub 2015 Dec 23. PMID 26701339
- [Background] Carter-Harris L, Brandzel S, Wernli KJ, Roth JA, Buist DSM. A qualitative study exploring why individuals opt out of lung cancer screening. Fam Pract. 2017 Apr 1;34(2):239-244. doi: 10.1093/fampra/cmw146. PMID 28122849
- [Background] Carter-Harris L, Slaven JE 2nd, Monahan PO, Draucker CB, Vode E, Rawl SM. Understanding lung cancer screening behaviour using path analysis. J Med Screen. 2020 Jun;27(2):105-112. doi: 10.1177/0969141319876961. Epub 2019 Sep 24. PMID 31550991
- [Background] Mohan G, Chattopadhyay S. Cost-effectiveness of Leveraging Social Determinants of Health to Improve Breast, Cervical, and Colorectal Cancer Screening: A Systematic Review. JAMA Oncol. 2020 Sep 1;6(9):1434-1444. doi: 10.1001/jamaoncol.2020.1460. PMID 32556187
- [Background] Weinstein D. The Precaution Adoption Process Model. In: Health Behavior and Health Education: Theory, Researchm and Practice. 4th Ed. Jossey-Bass; 2008:123-147.
- [Background] Chew LD, Bradley KA, Boyko EJ. Brief questions to identify patients with inadequate health literacy. Fam Med. 2004 Sep;36(8):588-94. PMID 15343421
- [Background] Thompson HS, Valdimarsdottir HB, Winkel G, Jandorf L, Redd W. The Group-Based Medical Mistrust Scale: psychometric properties and association with breast cancer screening. Prev Med. 2004 Feb;38(2):209-18. doi: 10.1016/j.ypmed.2003.09.041. PMID 14715214
- [Background] Cataldo JK, Slaughter R, Jahan TM, Pongquan VL, Hwang WJ. Measuring stigma in people with lung cancer: psychometric testing of the cataldo lung cancer stigma scale. Oncol Nurs Forum. 2011 Jan;38(1):E46-54. doi: 10.1188/11.ONF.E46-E54. PMID 21186151
- [Background] Mayo RM, Ureda JR, Parker VG. Importance of fatalism in understanding mammography screening in rural elderly women. J Women Aging. 2001;13(1):57-72. doi: 10.1300/J074v13n01_05. PMID 11217186
- [Background] Carter-Harris L, Slaven JE 2nd, Monohan P, Rawl SM. Development and Psychometric Evaluation of the Lung Cancer Screening Health Belief Scales. Cancer Nurs. 2017 May/Jun;40(3):237-244. doi: 10.1097/NCC.0000000000000386. PMID 27244666
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660